CLINICAL TRIAL: NCT00855712
Title: Prospective, Multicenter, Randomized, Clinical Investigation of TransMedics Organ Care System (OCS) for Cardiac Use
Brief Title: Randomized Study of Organ Care System Cardiac for Preservation of Donated Hearts for Eventual Transplantation
Acronym: PROCEEDII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TransMedics (Industry)
Collaborators: University of California, Los Angeles (Other); Columbia University (Other); The Cleveland Clinic (Other); Massachusetts General Hospital (Other); Newark Beth Israel Medical Center (Other); Cedars-Sinai Medical Center (Other); Groupe Hospitalier Pitie-Salpetriere (Other); Papworth Hospital NHS Foundation Trust (Other Government); Azienda Ospedaliera S. Maria della Misericordia (Other); Royal Brompton & Harefield NHS Foundation Trust (Other); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAR-05-2008
Record Dates: First submitted 2009-03-03; First posted 2009-03-04 (Estimated); Last update posted 2020-06-09 (Actual); Status verified 2015-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Transplant; Warm Perfusion; Organ Care; Resting Mode
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Organ Care System (Experimental)
  Interventions: Device: Organ Care System
- Cold cardioplegia solution (Active Comparator)
  Interventions: Device: Cold Cardioplegia Solution

INTERVENTIONS:
Device: Organ Care System — The Organ Care System (OCS) is a portable organ perfusion and monitoring system intended to preserve a donated heart in a near normal physiologic beating state during transport for eventual transplantation into a recipient. The OCS maintains organ viability by providing a controlled environment that simulates near-normal physiological conditions, continuously perfusing the donated heart with warm, oxygenated blood, supplemented with the Solution Set. The blood is collected from the donor and continuously circulated to the organ in a closed circuit along with the Solution. The OCS preserves and monitors the organ's perfusion and metabolic state after explantation from a donor and connection to the device, during transportation to the recipient site, and until disconnection from the device.
  Other Names: OCS
  Arms: Organ Care System
Device: Cold Cardioplegia Solution — This is the standard of care solutions used to arrest and preserve the donated heart during transport until arrival at recipient hospital
  Arms: Cold cardioplegia solution

SUMMARY:
The purpose of the study is to compare survival of both patients and newly transplanted hearts following heart transplantation among patients who were transplanted with donated hearts preserved on ice and those who were transplanted with donated hearts using the Organ Care System (OCS). The Organ care system preserves the hearts in a warm blood perfused beating state. The study also compares the number of rejection episodes, heart related adverse events, ICU time, and ventilation time between the two groups. The study is considered a success if survival in the OCS group was not inferior to the ice group.

ELIGIBILITY:
Inclusion Criteria:

Recipient Day of Transplant

* Registered male or female primary heart transplant candidate
* ≥18 years old
* Signed, written informed consent document and authorization to use and disclose protected health information

Donor Hearts

* <60 years old
* Mean systolic blood pressure >60 mmHg at the time of final heart assessment
* Satisfactory echocardiography assessment defined as:
* Ejection fraction >40%
* Absence of severe segmental wall motion abnormalities
* Absence of left ventricular hypertrophy (inter ventricular septum and posterior wall thickness <1.3 cm)
* Absence of valve abnormalities (trace to mild valvular regurgitation is acceptable)

Exclusion Criteria:

Recipient Day of Transplant

* >4 previous sternotomies
* Chronic renal failure as defined by chronic serum creatinine >3.0 mg/dL for more than 2 weeks and/or requiring hemodialysis (except for hemodialysis or hemofiltration for fluid overload)
* Ventilator dependence at the time of transplant
* Use of a ventricular assist device for > 30 days and the presence of any of the following: sepsis, intracranial hemorrhage or heparin induced thrombocytopenia
* Panel reactive antibodies > 40% with a positive prospective cross match and/or virtual cross match
* Use of an investigational drug or device, other than OCS, during the study.
* Simultaneous transplant of non-heart allograft, except for concurrent kidney transplant

Donor Hearts

* Abnormal coronary angiogram defined as >50% stenosis, requiring coronary bypass
* Donor-to-recipient body weight ratio of <0.6
* Inotrope support at time of final heart assessment including, but not limited to:

  * Dopamine >10 ug/kg/min
  * Dobutamine > 10 ug/kg/min
  * Milrinone >0.3 ug/kg/min
  * Epinephrine > 0.03 ug/kg/min
  * Norepinephrine > 0.03 ug/kg/min
  * Any bolus dose of the above prior to explants that would result in exceeding the above stated criteria
* Presence of any exclusion criterion based on the standard practice of the investigational site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-03; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
30-day patient survival following transplantation with the originally transplanted heart and no mechanical circulatory assist device at day 30 | 30 days

SECONDARY OUTCOMES:
Incidence of all cardiac graft-related serious adverse events | 30 days
Incidence of biopsy proven ISHLT grade 2R or 3R acute rejection on any of the surveillance endomyocardial biopsies or clinically symptomatic rejection requiring augmentation of immunosuppressive therapy during the 30 day follow up | 30 day
Length of ICU stay | 30 day

CONTACTS AND LOCATIONS:
Overall Officials: Abbas Ardehali, MD, Study Chair — University of California, Los Angeles
Locations (11):
- United States (7):
  - UCLA Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Columbia University Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
- Hospitalier Pitie-Salpetriere, Paris, France
- Azienda Ospedaliera S. Maria della Misericordia, Udine, Italy
- United Kingdom (2):
  - Papworth Hospital, Cambridge
  - Harefield Hospital, London

REFERENCES:
- [Derived] Ardehali A, Esmailian F, Deng M, Soltesz E, Hsich E, Naka Y, Mancini D, Camacho M, Zucker M, Leprince P, Padera R, Kobashigawa J; PROCEED II trial investigators. Ex-vivo perfusion of donor hearts for human heart transplantation (PROCEED II): a prospective, open-label, multicentre, randomised non-inferiority trial. Lancet. 2015 Jun 27;385(9987):2577-84. doi: 10.1016/S0140-6736(15)60261-6. Epub 2015 Apr 14. PMID 25888086